CLINICAL TRIAL: NCT04610619
Title: The Neuromuscular and Multisystem Features of RYR1-related Malignant Hyperthermia and Rhabdomyolysis - a Study Protocol
Brief Title: Multisystem Features of Malignant Hyperthermia or Rhabdomyolysis Related to RYR1 Variants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL72351.091.20
Record Dates: First submitted 2020-07-17; First posted 2020-10-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-07

CONDITIONS: Malignant Hyperthermia; Rhabdomyolysis; RYR1 Variant
MeSH Terms: conditions — Malignant Hyperthermia; Rhabdomyolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RYR1 related malignant hyperthermia/rhabdomyolysis
  Interventions: Other: Immunological challenge

INTERVENTIONS:
Other: Immunological challenge — In vitro immunological study of subjects with RYR1 related MH/rhabdomyolysis. Studying of circulating cytokines and cytokines production after in vitro stimulation

SUMMARY:
Rationale: Malignant hyperthermia and rhabdomyolysis are phenotypes that have long been considered to occur only in response to external stimuli (trigger anaesthesia and physical exhaustion) show several features of a continuous disease manifestation. Previous studies showed prolonged bleeding time after injury, selective immunological advantages, axial muscle weakness and several social difficulties. A detailed study of the neuromuscular and multisystem features of patients with RYR1-related malignant hyperthermia or rhabdomyolysis is needed to provide clarification about the continuous and multisystem disease manifestations in these patients.

Objective:

Primary Objective: There are three primary objectives in this study.

1. To investigate the neuromuscular involvement of RYR1 related MH and rhabdomyolysis.
2. To investigate the immunological changes in subjects with RYR1 related MH and rhabdomyolysis.
3. To identify multisystem features of RYR1 related MH and rhabdomyolysis.

There are no secondary objectives.

Study design: The design of the study will be a clinical, open, observational study. The study consists of three parts; a clinical, imaging and immunological part.

Study population: Patients with a history of malignant hyperthermia susceptibility (MHS), and/or a history of rhabdomyolysis related to a variant in RYR1.

Intervention (if applicable): Not applicable.

Main study parameters/endpoints: The study consists of three parts. Each part has it's own main study parameters

1. Clinical part: the results of the questionnaire study compared to standardizes normal values and the results of the comprehensive clinical assessment.
2. Imaging part: fatty infiltration and hypertrophy of proximal and axial muscles.
3. Immunological part: circulating and leukocyte released anti- and pro-inflammatory cytokine levels compared to healthy age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

* A history of malignant hyperthermia susceptibility (MHS), confirmed by diagnostic RYR1 variant or IVCT, related to a RYR1 variant and/or a history of rhabdomyolysis related to a variant in RYR1
* Minimum age 18 years old.

Exclusion Criteria:

* Patients diagnosed with a neuromuscular disease resulting in muscle weakness (apart from RYR1 related rhabdomyolysis and malignant hyperthermia).
* Patients with symptoms of angina pectoris.
* Patients with contra-indications for MRI-scan are excluded. Contra-indications for MRI-scan include metallic implants (vascular clips, foreign bodies like metallic splinters in the eye, coronary and peripheral artery stents, prosthetic heart valves, pacemakers and ICD's, cochlear implants, breast tissue expanders and some other electronic implants or devices and known claustrophobia.
* Current malignancy
* Pregnancy or lactating
* Other health issues whereby patients are not able to fulfil the study protocol
* No written informed consent by the patient

Exclusion criteria for immunological part of the study:

* Diabetes mellitus
* Patients currently using medicine affecting the immune system.
* Patients with a compromised immunity (e.g. HIV)• Patients with a history of auto-immune disease (e.g. SLE, psoriasis, IBD)
* Use of statins the past year
* Use of systemic corticosteroids during more than two weeks in the past 5 years
* Previous treatment with chemotherapy and/or radiation therapy
* Age > 65 years old.

Exclusion criteria for healthy controls

* History of malignant hyperthermia
* Variant in RYR1
* A RYR1 related myopathy
* History of heat stroke
* History of rhabdomyolysis
* Family history of malignant hyperthermia or a RYR1 variant
* Family history of inexplicable perioperative dead
* Family history of a RYR1 related myopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with RYR1 related malignant hyperthermia/rhabdomyolysis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the neuromuscular involvement of RYR1 related MH and rhabdomyolysis | Directly after inclusion, a muscle MRI's and ultra sounds will be made of all subjects.
  All subjects will have a total body muscle MRI and muscle ultra sound once
To investigate the multisystem features of RYR1 related MH and rhabdomyolysis | Directly after inclusion, subjects will fulfil a questionnaire study.
  All subject will fulfil a questionnaire study, it will focus on pain, activity and psychological aspects.
To investigate the multisystem features of RYR1 related MH and rhabdomyolysis | Six months after inclusion, subjects will fulfil a questionnaire study.
  All subject will fulfil a questionnaire study, it will focus on pain, activity and psychological aspects.
To investigate the multisystem features of RYR1 related MH and rhabdomyolysis | Twelve months after inclusion, subjects will fulfil a questionnaire study.
  All subject will fulfil a questionnaire study, it will focus on pain, activity and psychological aspects.
To investigate the immunological changes in subjects with RYR1 related MH and rhabdomyolysis. | Directly after inclusion blood samples will be taken for immunological studies.
  Peripheral mononuclear blood cells will be isolated and in vitro challenged using pathogens and stimulatia. The results of this part of the study will be compared to healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- RUniversity, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be shared with other researchers
Supporting Information: Study Protocol

REFERENCES:
- [Derived] van den Bersselaar LR, Kruijt N, Scheffer GJ, van Eijk L, Malagon I, Buckens S, Custers JA, Helder L, Greco A, Joosten LA, van Engelen BG, van Alfen N, Riazi S, Treves S, Jungbluth H, Snoeck MM, Voermans NC. The neuromuscular and multisystem features of RYR1-related malignant hyperthermia and rhabdomyolysis: A study protocol. Medicine (Baltimore). 2021 Aug 20;100(33):e26999. doi: 10.1097/MD.0000000000026999. PMID 34414986